CLINICAL TRIAL: NCT04521062
Title: Dilapan-S® for Induction of Labor - Assessing ouTpatient Placement and Effectiveness - The Feasibility Study (The DILATE Study).
Brief Title: Dilapan-S® for Induction of Labor The Feasibility Study
Acronym: DILATE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low recruitment
Sponsor: Albany Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 5768
Record Dates: First submitted 2020-07-07; First posted 2020-08-20 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Induction of Labor Affected Fetus / Newborn
Keywords: cervical ripening; induction of labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Dilapan S (Other): Placement of dilators
  Interventions: Device: Dilapan S

INTERVENTIONS:
Device: Dilapan S — Placement of Dilapan S

SUMMARY:
This is a prospective feasibility study to investigate Dilapan-S® as an outpatient method of cervical ripening in low risk pregnancies >=39 weeks.

DETAILED DESCRIPTION:
In 2019, the ARRIVE trial was published, demonstrating that in low risk nulliparous women, induction of labor at 39 weeks was associated with a decreased risk for hypertensive disorders of pregnancy and decreased risk for cesarean without any increased risk for severe neonatal complications or perinatal death. (1) Based on the results of this trial, hospitals have been questioning the feasibility of implementing a protocol which offers induction of labor to low risk women at ≥39 weeks. There are concerns regarding the ability of a busy labor and delivery to accommodate women presenting for inductions with an unfavorable cervix. Outpatient mechanical cervical ripening would allow for women to start the process of induction of labor at home. This is appealing because cervical ripening is typically the longest component of the induction process. Mechanical cervical ripening is the process by which balloons or dilators are placed into the cervix.

There is lack of evidence on Dilapan-S® as an outpatient method of cervical ripening despite the potential benefits of increased maternal satisfaction and decreased length of hospital stay. With this in mind we propose a preliminary study of 40 women to assess for feasibility of performing a large randomized control trial and assess safety with outpatient treatment. This initial study is intended to assess the feasibility of outpatient cervical ripening, next day induction of labor, and safety. After completion of this feasibility study, the investigators plan to initiate a randomized control trial to assess the efficacy of outpatient Dilapan-S® for mechanical cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

1. Planned induction of labor ≥ 39 weeks
2. Singleton gestation
3. Vertex presentation
4. Cervical dilation <3cm

Exclusion Criteria:

1. Placenta previa
2. Placenta accreta
3. Vasa previa
4. Preterm prelabor rupture of membranes
5. Non-english speaking
6. <18 years old
7. Multiple gestation
8. Prior cesarean delivery
9. Prior myomectomy
10. Fetal malpresentation
11. Active vaginal bleeding
12. Cervical dilation >1 cm
13. Uterine anomaly (didelphysis, bicornuate)
14. Intrauterine growth restriction <10th%
15. Fetal anomalies
16. Requirements to be inpatient
17. Polyhydramnios (AFI>25cm or MVP>8cm)
18. Chronic hypertension on medications
19. Gestational hypertension/preeclampsia
20. GDMA2, DM1, DM2
21. Hepatitis B or C
22. HIV

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Time to delivery | from induction start to delivery, estimated average 12 hours
  Length of time between induction of labor start and delivery (hours)

SECONDARY OUTCOMES:
APGAR score at 1and 5 min | 1 and 5 minutes after birth
  APGAR score (number 0-10)
number of participants with maternal infection | during hospital admission, average 4 days
  chorioamnionitis, endometritis - Yes/No
NICU admission | through maternal hospital admission, average 4 days
  Neonatal admission to NICU (any admission) - Yes/No
Need for neonatal antibiotics | in the first 72 hours after delivery
  any antibiotic use in postnatal period (yes/no)
Need for resipiratory support | during hospital admission, average 4 days
  any respiratory interventions after birth for neonate (composite of oxygen administration, respiratory distress syndrome, CPAP, intubation) (yes/No)
mode of delivery | one time at the time of delivery, variable to occur during hospital admission, average 4 days
  cesarean or vaginal (coded as cesarean delivery Y/N or vaginal delivery Y/N)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lynch, MD, Principal Investigator — Albany Medical College
Locations (1):
- Albany Medical Center, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No